CLINICAL TRIAL: NCT06611462
Title: Effect of Tailored, Intensive Prehabilitation for Risky Lifestyles Before Ventral Hernia Repair on Postoperative Outcomes, Health, and Costs - a Randomised Controlled Trial (STRONG-Hernia)
Brief Title: STRONG for Surgery & Strong for Life - Intensive Prehabilitation for Risk Reduction in Ventral Hernia Repair
Acronym: STRONG-Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Zealand University Hospital (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Hanne Tonnesen, Clinical Professor, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-23028872
Record Dates: First submitted 2024-02-13; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Ventral Hernia; Surgery; Risk Reduction; Lifestyle; Postoperative Complications; Prehabilitation
Keywords: Ventral Hernia; Surgery; Risk Reduction; Postoperative Complications; Prehabilitation; Smoking; Alcohol drinking; Obesity; Malnutrition; Physical Inactivity
MeSH Terms: conditions — Hernia, Ventral; Risk Reduction Behavior; Postoperative Complications; Smoking; Alcohol Drinking; Obesity; Malnutrition; Sedentary Behavior | interventions — Preoperative Exercise; Ethanol; Exercise; Nutritional Support

STUDY DESIGN:
Intervention Model Description: Randomised parallel design using block randomisation. Stratification for centre and number of SNAP factors (one, two, or ≥ 3).
Masking Description: Statistical analyses will be conducted blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation (Experimental): Intervention (the STRONG programme): At least six counselling sessions (around one per week) prior to surgery as an integrated prehabilitation programme tailored to the individual patient's need for risk reduction at surgery based on a baseline screening for risky SNAP factors. It is delivered via the surgical "Engage in the process of change". The smoking cessation intervention follows the Gold Standard Programme and a similar structure has been used for alcohol cessation, physical exercise, and nutrition interventions. All participants in the intervention group will receive immunonutrition in the days before surgery.
  Interventions: Behavioral: Prehabilitation (the STRONG programme)
- Treatment as usual (No Intervention): Treatment as usual in the preoperative period in the included hospital departments, e.g. brief counselling/advice regarding smoking cessation and weight loss, and handing out the national folders on smoking and surgery. Participants are free to access support to lifestyle changes in the community.

INTERVENTIONS:
Behavioral: Prehabilitation (the STRONG programme) — Participants screened positive for one or more SNAP factors and randomised to the intervention group will receive an individualised plan for prehabilitation of their specific SNAP factors.
  Other Names: Smoking cessation; Alcohol cessation; Physical activity; Nutritional support for malnutrition and/or obesity
  Arms: Prehabilitation

SUMMARY:
The five risky lifestyles Smoking, Nutrition (obesity and malnutrition), risky Alcohol intake, and Physical inactivity (SNAP) are common in surgical patients and associated with worse postoperative outcomes. Mono-factor interventions targeting and improving these risky lifestyles have been shown to reduce the risk at surgery, but there is a lack of systematic assessment of all five lifestyles of the patient before surgery and related optimization.

This study aims to evaluate the effect of intensive combined lifestyle interventions (the STRONG programme) compared with treatment as usual in patients undergoing ventral hernia repair on postoperative complications, health, and costs on short and longer term.

The hypothesis is that the STRONG programme will halve the complication rates within 30 days.

DETAILED DESCRIPTION:
This study is a multicentre randomised controlled trial. A total of 400 participants with one or more of the five risky SNAP lifestyles will be randomised to either the STRONG programme (a prehabilitation intervention) or treatment as usual preoperatively (control). The STRONG programme is individually tailored to the needs of the participants. The program contains education, motivational, and pharmaceutical support. All participants will be followed up at the end of the intervention/at surgery, one, three, and six months after surgery. Long-term outcomes are followed up from national registers two years after surgery.

Interim analysis will be employed.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years scheduled for ventral hernia repair (defect smaller than 8cm)
* Enough time for at least 4 weeks of prehabilitation
* Screened positive for at least 1 risky SNAP factor
* Signed informed consent

Exclusion Criteria:

* Ventral hernia repairs with defect larger than 8 cm
* Pregnancy/breastfeeding
* Allergy/other contradiction to pharmaceutical and/or nutritional support
* Contradiction to exercise
* Previous complicated alcohol withdrawal symptoms (delirium or seizures)
* Not able to participate in intervention due to psychiatric ilness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications within 30 days | 30 days
  Number and proportion of participants with at least one postoperative complication defined by requiring treatment

SECONDARY OUTCOMES:
Postoperative complications within 3 and 6 months | 3 months, 6 months
  Number and proportion of participants with at least one postoperative complication defined by requiring treatment
Comprehensive Complication Index (CCI) | 30 days, 3 months, 6 months
  Calculated from the Clavien-Dindo classification of the postoperative complications
Successful quitting of risky lifestyles | End of intervention/at surgery, 30 days, 3 months, 6 months
  Number and proportion of participants without all of their preoperative risky lifestyles (identified at baseline). Successful quitting of risky lifestyles are defined as:
  * Smoking: no use of any tobacco products
  * Malnutrition: not at risk of malnutrition defined as NRS <3
  * Obesity: 5-10 % loss of body fat mass compared to baseline
  * Alcohol: Zero alcohol intake at end of intervention/surgery and below risky limits (<14 units per week) at postoperative follow-ups
  * Physical inactivity: being physically active at least 3.5 hours per week
Any improvement of risky lifestyles | End of intervention/at surgery, 30 days, 3 months, 6 months
  Number and proportion of participants with any improvement of any of their risky lifestyles compared with baseline. Any improvements include:
  * Smoking: a reduced number of cigarettes
  * Malnutrition: improvement in level of malnutrition (NRS scale)
  * Obesity: any loss of body fat mass
  * Alcohol: a reduced alcohol intake weekly (reduced number of units weekly)
  * Physical inactivity: Any improvement in minutes of daily physical activity
Health-Related Quality of Life (HRQoL) | End of intervention/at surgery, 30 days, 3 months, 6 months
  Number and proportion of patients with improvement of HRQoL compared with baseline. HRQoL is measured by the EQ-5D instrument
Costs | 30 days, 6 months, 2 years
  Measured as individual direct and indirect healthcare costs per patient based on data from national registries
Cost-effectiveness | 2 years
  Calculated as a probability in percent (%)
Patient expectations | Baseline
  Measured as a number on a VAS scale from 0-10
Patient reflections 1 | Baseline
  Qualitative analysis of patients reflections on advantages and disadvantages of changing or continuing current lifestyle
Patient reflections 2 | Baseline
  Qualitative analysis of patient reflections obtained from semi-structured interviews

OTHER OUTCOMES:
Postoperative length of stay | From surgery until 30 days postoperative
  Descriptively reported as total time in hospital within 30 postoperative days with 95% CI
Readmission | 90 days
  Descriptively reported as number and proportion (in %) of participants with readmission with 95% CI
Time back to work/usual activities | 30 days, 3 months, 6 months
  Descriptively reported, patient reported
Hernia recurrence | 90 days
  Descriptively reported as number and proportion of participants with hernia recurrence
Reoperation for hernia recurrence | 90 days
  Descriptively reported as number and proportion (in %) of participants reoperated for hernia recurrence with 95% CI
Visits to primary care | 30 days
  Descriptively reported as number and proportion (in %) of participants with any visits to primary care with 95% CI
Successful quitting of risky lifestyles individually | End of intervention/at surgery, 30 days, 3 months, 6 months
  Descriptively reported as number and proportion (in%) of participants without their preoperative risky lifestyle (identified at baseline) with 95% CI. Each lifestyle is reported separately. Successful quitting of risky lifestyles are defined as:
  * Smoking: no use of any tobacco products
  * Malnutrition: not at risk of malnutrition defined as NRS <3
  * Obesity: 5-10 % loss of body fat mass compared to baseline
  * Alcohol: Zero alcohol intake at end of intervention/surgery and below risky limits (<14 units per week) at postoperative follow-ups
  * Physical inactivity: being physically active at least 3.5 hours per week
Change in ASA score | End of intervention/at surgery, 30 days, 3 months, 6 months
  Descriptively reported as number and proportion (in %) of participants with change in ASA score level compared with baseline related to a change in risky SNAP factors with 95% CI
Change of frailty | End of intervention/at surgery, 30 days, 3 months, 6 months
  Descriptively reported as number and proportion (in %) of participants with change in frailty score compared with baseline with 95% CI. Measured by Fried's Modified Frailty Score.
Morbidity | 2 years
  Descriptively reported as grouped diagnoses via the Danish version of ICD-10 based on data from the Danish National Patient Registry.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, Professor MD, Principal Investigator — WHOCC, The Parker Institute, Bispebjerg-Frederiksberg Hospital, RegH, Copenhagen
Locations (3):
- Denmark (3):
  - Copenhagen University Hospital at Herlev, Herlev
  - Holbaek Sygehus, Holbæk
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen SAS, Lauridsen SV, Fonnes S, Rosenberg J, Tonnesen H. Effect of tailored, intensive prehabilitation for risky lifestyles before ventral hernia repair on postoperative outcomes, health, and costs - study protocol for a randomised controlled trial (STRONG-Hernia). PLoS One. 2025 May 28;20(5):e0324002. doi: 10.1371/journal.pone.0324002. eCollection 2025. PMID 40435308